CLINICAL TRIAL: NCT02144285
Title: A Single-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3113593 in Healthy Subjects and Patients With Chronic Kidney Disease Treated With Hemodialysis
Brief Title: A Study of LY3113593 in Healthy Participants and Participants With Chronic Kidney Disease Treated With Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 15200; I7C-MC-FEAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2018-08

CONDITIONS: Kidney Failure, Chronic
Keywords: Renal dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- LY3113593 IV (Part A) (Experimental): Single dose of LY3113593 administered intravenous (IV) at a minimum of six dose levels
  Interventions: Drug: LY3113593
- Placebo IV (Part A) (Placebo Comparator): Single dose of placebo matching LY3113593 administered IV
  Interventions: Drug: Placebo
- LY3113593 SC (Part A) (Experimental): Single dose of LY3113593 administered subcutaneous (SC)
  Interventions: Drug: LY3113593
- Placebo SC (Part A) (Placebo Comparator): Single dose of placebo matching LY3113593 administered SC
  Interventions: Drug: Placebo
- LY3113593 IV (Part B) (Experimental): Single dose of LY3113593 administered IV
  Interventions: Drug: LY3113593
- Placebo IV (Part B) (Placebo Comparator): Single dose of placebo matching LY3113593 administered IV
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3113593 — Administered IV
  Arms: LY3113593 IV (Part A); LY3113593 IV (Part B)
Drug: LY3113593 — Administered SC
  Arms: LY3113593 SC (Part A)
Drug: Placebo — Administered IV
  Arms: Placebo IV (Part A); Placebo IV (Part B)
Drug: Placebo — Administered SC
  Arms: Placebo SC (Part A)

SUMMARY:
The purpose of this study is to look at the tolerability and safety of LY3113593. Study doctors will see how safe it is and whether it produces side effects following a single injection into a vein or under the skin in healthy participants (Part A) and participants with chronic kidney disease treated with hemodialysis (Part B). The study will also measure how much of the study drug gets into the blood stream, how long it takes the body to get rid of the study drug and what effects the study drug has on the body.

This is the first time that this study drug is being given to participants. This study is for research purposes only and is not intended to treat any medical condition. For each participant, the study will last about 85 days, not including screening. Screening is required within 28 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Participants:

  * Healthy males or females
  * Participants have a body mass index (BMI) of 18.5 to 29.9 kilogram per meter square (kg/m^2), inclusive at screening
* Participants Treated with Hemodialysis:

  * Participants are males or females who have end-stage renal disease (ESRD) and have been receiving adequate maintenance hemodialysis (3 times weekly) for at least 12 weeks prior to screening
  * Participants have a hemoglobin value greater than or equal to (≥)9.0 grams per deciliter (g/dL) and less than or equal to (≤)12.5 g/dL at screening
  * Participants have a body mass index (BMI) of 18.5 to 45.0 kg/m^2, inclusive, at screening
* Both Populations:

  * Male participants agree to use a reliable method of birth control and avoid donating sperm during the study and for 3 months following the dose of the investigational product
  * Female participants must not be of child-bearing potential

Exclusion Criteria:

* Healthy Participants:

  * Participants that have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
  * Participants that have used or intend to use over-the-counter or prescription medication, including herbal medications within 14 days prior to dosing
* Participants Treated with Hemodialysis:

  * Participants that have a history of myocardial infarction, acute coronary syndrome, stroke or transient ischemic attacks within the prior 6 months
  * Participants that have heart failure that results in dyspnea at rest or during minimal exercise
  * Participants that have poorly controlled hypertension
  * Participants that have a history of significant thrombotic disease, pulmonary hypertension, significant hematological disease or current liver disease, known hepatic or biliary abnormalities
  * Participants that had a blood transfusion within the prior 12 weeks or an anticipated need for blood transfusion during the study
  * Participants that have evidence of active peptic, duodenal, or esophageal ulcer disease or gastrointestinal bleeding within the prior 12 weeks
* Both Populations:

  * Participants that have known allergies to related compounds or any components of the study drug or its formulation, clinically significant multiple or severe drug allergies, or intolerance to topical corticosteroids, or severe post treatment hypersensitivity reactions or history of significant atopy
  * Participants that have participated, within the last 30 days (or 5 half-lives if long half life) in a clinical trial involving an investigational product
  * Participants that have known or ongoing psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Parexel Early Phase Unit at Glendale, Glendale, California
  - Orlando Clinical Research Center, Orlando, Florida
  - Davita Clinical Research, Minneapolis, Minnesota

REFERENCES:
- [Derived] Sheetz M, Barrington P, Callies S, Berg PH, McColm J, Marbury T, Decker B, Dyas GL, Truhlar SME, Benschop R, Leung D, Berg J, Witcher DR. Targeting the hepcidin-ferroportin pathway in anaemia of chronic kidney disease. Br J Clin Pharmacol. 2019 May;85(5):935-948. doi: 10.1111/bcp.13877. Epub 2019 Mar 4. PMID 30677788

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Part A): Single dose of placebo matching LY3113593.
- LY IV 1.5mg (Part A): Single dose of LY3113593 (LY) administered IV at a 1.5 milligrams (mg).
- LY IV 5mg (Part A): Single dose of LY3113593 administered intravenous (IV) at 5 mg.
- LY IV 15mg (Part A): Single dose of LY3113593 administered IV at 15 mg.
- LY IV 50mg (Part A): Single dose of LY3113593 administered IV at 50 mg.
- LY IV 150mg (Part A); LY IV 150mg(Part B): Single dose of LY3113593 administered IV at 150 mg.
- LY IV 400mg (Part A): Single dose of LY3113593 administered IV at 400 mg.
- LY SC 150mg (Part A): Single dose of LY3113593 administered subcutaneously (SC) at 150 mg.
Period: Overall Study
Arm/Group | Placebo (Part A) | LY IV 1.5mg (Part A) | LY IV 5mg (Part A) | LY IV 15mg (Part A) | LY IV 50mg (Part A) | LY IV 150mg (Part A) | LY IV 400mg (Part A) | LY SC 150mg (Part A) | Placebo IV (Part B) | LY IV 150mg(Part B)
Started | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 6
Received At Least One Dose of Study Drug | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 6
Completed | 14 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 2 | 6
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- LY IV 150mg (Part B): Single dose of LY3113593 administered IV at 150 mg.
- Total: Total of all reporting groups
Arm/Group | Placebo (Part A) | LY IV 1.5mg (Part A) | LY IV 5mg (Part A) | LY IV 15mg (Part A) | LY IV 50mg (Part A) | LY IV 150mg (Part A) | LY IV 400mg (Part A) | LY SC 150mg (Part A) | Placebo IV (Part B) | LY IV 150mg (Part B) | Total
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 6 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All enrolled participants Age data as per Part in trial.
  years
    Part A: number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 56
    Part A | 37.8 (10.69) | 45.0 (7.40) | 31.0 (5.22) | 30.7 (4.41) | 41.5 (21.00) | 46.3 (8.89) | 38.3 (7.55) | 43.7 (13.05) |  |  | 39.1 (11.49)
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6 | 8
    Part B |  |  |  |  |  |  |  |  | 38.5 (13.44) | 51.7 (5.85) | 48.4 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 2 | 9
  Male | 13 | 4 | 6 | 6 | 6 | 2 | 6 | 6 | 2 | 4 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 1 | 0 | 1 | 1 | 0 | 3 | 1 | 0 | 13
  Not Hispanic or Latino | 12 | 2 | 5 | 6 | 5 | 5 | 6 | 3 | 1 | 6 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 0 | 0 | 3 | 3 | 3 | 0 | 0 | 0 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 6 | 3 | 0 | 1 | 1 | 0 | 0 | 6 | 22
  White | 7 | 4 | 0 | 3 | 3 | 1 | 2 | 6 | 2 | 0 | 28
  More than one race | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 6 | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event (s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: The number of participants with 1 or more SAEs assessed as related to the study drug and is summarized cumulatively. A serious adverse event is defined as an event that results in death, initial or prolonged hospitalization, is life-threatening, leads to persistent or significant disability/incapacity, is associated with congenital anomaly/birth defect, or is considered significant by the investigator for any other reason. A summary of all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline through end of study (Day 85)
Population: All enrolled participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo IV (Part B): Single dose of LY3113593 administered IV.
Arm/Group | Placebo (Part A) | LY IV 1.5mg (Part A) | LY IV 5mg (Part A) | LY IV 15mg (Part A) | LY IV 50mg (Part A) | LY IV 150mg (Part A) | LY IV 400mg (Part A) | LY SC 150mg (Part A) | Placebo IV (Part B) | LY IV 150mg (Part B)
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY3113593
Time Frame: Day 1: pre-dose, 30 minutes, 2 hours, 4 hours, 12 hours; Days 2, 3, 5, 8, 15, 22, 29, 43, 57, 71, and 85
Population: All enrolled participants who received at least one dose of LY3113593 study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- LY SC 150 mg (Part A): Single dose of LY3113593 administered subcutaneously (SC) at 150 mg.
- LY IV 150 mg (Part B): Single dose of LY3113593 administered IV at 150mg.
Arm/Group | LY IV 1.5mg (Part A) | LY IV 5mg (Part A) | LY IV 15mg (Part A) | LY IV 50mg (Part A) | LY IV 150mg (Part A) | LY IV 400mg (Part A) | LY SC 150 mg (Part A) | LY IV 150 mg (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanograms per milliliter (ng/mL) | 559 (15) | 2070 (14) | 6330 (13) | 20000 (19) | 60800 (34) | 170000 (13) | 11300 (43) | 38000 (31)

3. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve to Infinity (AUC (0-∞)) of LY3113593
Time Frame: Day 1: pre-dose, 30 minutes, 2 hours, 4 hours, 12 hours; Days 2, 3, 5, 8, 15, 22, 29, 43, 57, 71, and 85
Population: All enrolled participants who received at least one dose of LY3113593 study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | LY IV 1.5mg (Part A) | LY IV 5mg (Part A) | LY IV 15mg (Part A) | LY IV 50mg (Part A) | LY IV 150mg (Part A) | LY IV 400mg (Part A) | LY SC 150 mg (Part A) | LY IV 150mg (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanograms*hour per milliliter (ng*hr/mL) | 55700 (29) | 280000 (14) | 1100000 (9) | 5240000 (17) | 17000000 (28) | 38300000 (17) | 7640000 (37) | 8270000 (34)

4. Secondary Outcome: Pharmacokinetics: Absolute Bioavailability of LY3113593 SC Versus IV Based on AUC Ratios
Time Frame: Day 1: pre-dose, 30 minutes, 2 hours, 4 hours, 12 hours; Days 2, 3, 5, 8, 15, 22, 29, 43, 57, 71, and 85
Population: All enrolled participants who received at least one dose of 150mg LY3113593 study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- LY IV 150mg (Part A): Single dose of LY3113593 (LY) administered IV at 150 mg.
Arm/Group | LY SC 150mg (Part A) | LY IV 150mg (Part A)
Number analyzed (Participants) | 6 | 6
ng*h/mL | 7640000 (37) | 17000000 (28)
Statistical Analysis 1: Comparison: LY SC 150mg (Part A) vs LY IV 150mg (Part A); Test type: Superiority or Other; Absolute Bioavailability = 0.45, 90% CI 2-sided [0.34 to 0.60]

5. Secondary Outcome: Pharmacodynamics: Maximum Change From Baseline in Iron Parameter Profile of LY3113593
Time Frame: Baseline, Day 85
Population: All enrolled participants who received at least one dose of study drug and had baseline and post baseline iron profile data.
Measure: Mean (Standard Deviation); unit: micromoles per liter (μmol/L)
Groups:
- LY IV (Part B): Single dose of LY3113593 administered IV.
Arm/Group | Placebo (Part A) | LY IV 1.5mg (Part A) | LY IV 5mg (Part A) | LY IV 15mg (Part A) | LY IV 50mg (Part A) | LY IV 150mg (Part A) | LY IV 400mg (Part A) | LY SC 150mg (Part A) | Placebo IV (Part B) | LY IV (Part B)
Number analyzed (Participants) | 12 | 6 | 5 | 6 | 6 | 6 | 5 | 6 | 2 | 6
micromoles per liter (μmol/L) | 6.78 (12.5) | 4.12 (5.49) | 9.46 (11.6) | 8.38 (5.22) | 10.23 (10.8) | 13.5 (5.68) | 7.9 (9.67) | 6.97 (14.4) | 3.3 (1.98) | 7.92 (6.68)

6. Secondary Outcome: Pharmacodynamics: Maximum Absolute Change From Baseline in TSat Parameter Profile of LY3113593
Time Frame: Baseline, Day 85
Population: All enrolled participants who received at least one dose of study drug and had baseline and post baseline Tsat profile data.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Placebo (Part A) | LY IV 1.5mg (Part A) | LY IV 5mg (Part A) | LY IV 15mg (Part A) | LY IV 50mg (Part A) | LY IV 150mg (Part A) | LY IV 400mg (Part A) | LY SC 150mg (Part A) | Placebo IV (Part B) | LY IV (Part B)
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 2 | 6
percentage of change | 11.00 (22.00) | 6.80 (10.00) | 14.80 (18.00) | 15.70 (11.00) | 12.80 (23.00) | 21.00 (8.60) | 07.80 (6.65) | 17.00 (16.00) | -0.50 (14.90) | 18.30 (18.10)

7. Secondary Outcome: Pharmacodynamics: Maximum Change From Baseline in Hemoglobin (Hb) Parameter Profile of LY3113593
Time Frame: Baseline, Day 85
Population: All enrolled participants who received at least one dose of study drug and had baseline and post baseline Hb profile data.
Measure: Mean (Standard Deviation); unit: millimoles per liter of iron (mml/L-Fe)
Arm/Group | Placebo (Part A) | LY IV 1.5mg (Part A) | LY IV 5mg (Part A) | LY IV 15mg (Part A) | LY IV 50mg (Part A) | LY IV 150mg (Part A) | LY IV 400mg (Part A) | LY SC 150mg (Part A) | Placebo IV (Part B) | LY IV (Part B)
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 5 | 6 | 6 | 5 | 2 | 6
millimoles per liter of iron (mml/L-Fe) | 0.269 (0.455) | 0.425 (0.363) | 0.123 (0.486) | 0.205 (0.468) | 0.780 (0.38) | 0.508 (0.65) | 0.165 (0.796) | 0.217 (0.306) | 0.375 (0.361) | 0.568 (0.444)

ADVERSE EVENTS:
Description: All enrolled participants.
Arm/Group | Placebo (Part A) | LY IV 1.5mg (Part A) | LY IV 5mg (Part A) | LY IV 15mg (Part A) | LY IV 50mg (Part A) | LY IV 150mg (Part A) | LY IV 400mg (Part A) | LY SC 150mg (Part A) | Placebo IV (Part B) | LY IV (Part B)
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 1/6
Other Adverse Events (participants affected / at risk) | 4/14 | 3/6 | 2/6 | 2/6 | 5/6 | 3/6 | 2/6 | 2/6 | 0/2 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=14) | LY IV 1.5mg (Part A) (N=6) | LY IV 5mg (Part A) (N=6) | LY IV 15mg (Part A) (N=6) | LY IV 50mg (Part A) (N=6) | LY IV 150mg (Part A) (N=6) | LY IV 400mg (Part A) (N=6) | LY SC 150mg (Part A) (N=6) | Placebo IV (Part B) (N=2) | LY IV (Part B) (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=14) | LY IV 1.5mg (Part A) (N=6) | LY IV 5mg (Part A) (N=6) | LY IV 15mg (Part A) (N=6) | LY IV 50mg (Part A) (N=6) | LY IV 150mg (Part A) (N=6) | LY IV 400mg (Part A) (N=6) | LY SC 150mg (Part A) (N=6) | Placebo IV (Part B) (N=2) | LY IV (Part B) (N=6)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days